CLINICAL TRIAL: NCT05530850
Title: The Effect of Holistic Corrective Exercise Program on Kyphosis Degree, Balance and Quality of Life in Kyphotic Adolescent
Brief Title: The Effect of Holistic Corrective Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Doctor Of Philosophy, Hasan Kalyoncu University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HKU-GE-KYPHOSİS
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Kyphosis Thoracic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Holistic Corrective Exercise Program (Experimental): A holistic approach corrective exercise program including corrective exercises and postural perception training
  Interventions: Behavioral: Holistic Corrective Exercise Program
- Thoracic exercise program (Experimental): Thoracic region focused exercise program
  Interventions: Other: Thoracic exercise program
- control group (No Intervention): Individuals in the control group were asked to continue their activities of daily living.

INTERVENTIONS:
Behavioral: Holistic Corrective Exercise Program — A holistic approach corrective exercise program including corrective exercises and postural perception training,
  Arms: Holistic Corrective Exercise Program
Other: Thoracic exercise program — Thoracic region focused exercise program
  Arms: Thoracic exercise program

SUMMARY:
This study was planned to investigate the effect of holistic approach corrective exercise program on the degree of kyphosis, balance and quality of life in kyphotic adolescents. A holistic approach corrective exercise program including corrective exercises and postural perception training was applied to one group. Thoracic region focused exercise program was applied to the other group. The programs of the exercise groups were applied three days a week, for 12 weeks. The kyphosis angle of all individuals participating in the study was evaluated using the flexible ruler, the Romberg index measured with balance pedobarography, and the quality of life using the Scoliosis Research Society-22 Questionnaire (SRS-22). In our study, a decrease in the degree of kyphosis was detected in the holistic approach corrective exercise and thoracic region-focused exercise group after 12 weeks of exercise training (p<0.001), while no change was observed in the control group (p>0.05). Balance improved after exercise training in the holistic corrective exercise group (p=0.006). The quality of life increased in the holistic approach corrective exercise and thoracic region focused exercise groups after the training (p<0.001). The use of postural perception training together with corrective exercise programs in applications for thoracic kyphosis reveals a holistic approach and may increase the effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male individual between the ages of 10-18,
* Kyphosis degree ≥50°,

Exclusion Criteria:

* Rrigid thoracic kyphosis
* Scoliosis with a Cobb angle >10°
* Congenital spine problem,
* Shoulder, pelvis and other spinal injuries

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
The Kyphosis angle by using flexible ruler | 12 weeks
  Flexible ruler

SECONDARY OUTCOMES:
Balance assesment by using the romberg index | 12 weeks
  the Romberg index, Pedobarography

OTHER OUTCOMES:
Quality of Life by using SRS-22 | 12 weeks
  Scoliosis Research Society-22 Questionnaire (SRS-22)

CONTACTS AND LOCATIONS:
Overall Officials: GÖNÜL ELPEZE, Principal Investigator — HKU
Locations (1):
- Hasan Kalyoncu Üniversitesi, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No